CLINICAL TRIAL: NCT03853564
Title: Clinical Trial of an Early Parenting Empowerment Intervention to Promote Socioemotional Development in Infants With Developmental Disabilities: Parent and Infant Behavioral, Neuroendocrine and Epigenetics Outcomes
Brief Title: Early Parenting Intervention: Bio-behavioral Outcomes in Infants With Neurodevelopmental Disabilities
Acronym: EPI-BOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Fondazione Istituto Neurologico Casimiro Mondino (Unknown); Università degli Studi di Brescia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RF-2016-02361884
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Epigenomics; Developmental Disability; Early Intervention; Parent-Child Relations
Keywords: DNA methylation; Epigenetic regulation; Video-feedback intervention; Developmental disability; Cerebral palsy; Genetic syndromes; Parent-infant interaction; Early intervention; Neuroendocrine regulation
MeSH Terms: conditions — Developmental Disabilities; Cerebral Palsy; Genetic Diseases, Inborn

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-Feedback Group (VFG) (Experimental): Dyads of mothers and their infant with developmental disability who are exposed to the video-feedback intervention focused on different domains of mother-infant quality of interaction (number of sessions: 6).
  Interventions: Behavioral: Video-Feedback Intervention
- Phone-Call Group (PCG) (Sham Comparator): Dyads of mothers and their infant with developmental disability who are not exposed to the video-feedback intervention, instead they receive phone calls focused on obtaining descriptions of different domains of infant behavioral development (number of sessions: 6)
  Interventions: Other: Phone-Call Intervention

INTERVENTIONS:
Behavioral: Video-Feedback Intervention — Mothers and infants of the VFG arm will participate to a 6-session video-feedback intervention structured as follows: 4 sessions of video-review discussions with a trained clinician + 2 sessions of integrative intervention aimed at translating into practical caregiving the insights developed during the video-review discussions.
  Arms: Video-Feedback Group (VFG)
Other: Phone-Call Intervention — Mothers of the PCG arm will participate in 6-session of telephone call during which a trained collaborator will ask details on different domains of infants behavioral development.
  Arms: Phone-Call Group (PCG)

SUMMARY:
Infants with developmental disabilities present a high risk of behavioral and socio-emotional problems. Their parents are themselves at risk of developing emotional and affective disorders which can impact the quality of the interaction with the infant. Early parenting empowerment focused on parent-infant interaction are beneficial in supporting infants development and parental adjustment. By using a multi-layer approach to outcomes assessment (i.e., behavioral, neuroendocrine and epigenetic outcomes), the present longitudinal, multi-center, change-promoting clinical trial is aimed at assessing the effectiveness of an early parenting empowerment intervention based on video-feedback technique to support maternal responsiveness and the socio-emotional development of infants with developmental disabilities.

DETAILED DESCRIPTION:
RATIONALE: Infants with developmental disabilities (e.g., cerebral palsy and genetic syndrome) present a high risk of behavioral and socio-emotional problems. Their parents are themselves at risk of developing emotional and affective disorders which can impact the quality of the interaction with the infant. Typical development research is highlighting the potentials of biological markers of less-than-optimal mother-infant interaction, such as altered neuroendocrine regulation (i.e., cortisol and oxytocin). Increased infants' salivary cortisol reactivity has been found in response to experimental suspension of maternal responsiveness (Still-Face paradigm, SFP). On the other hand, oxytocin administration to mothers increases responsiveness to infants socio-emotional signals and oxytocin has also been associated with socioemotional stress regulation in humans. Interestingly, previous research suggests that the epigenetic regulation of specific genes (i.e., SLC6A4, NR3C1, BDNF, OXTR) transcription might be affected by alterations of maternal caregiving behavior. Nonetheless, to the best of our knowledge, to date there is no investigation of the epigenetic vestiges of the effects of an early parenting intervention (i.e., video-feedback) on the behavioral outcomes of infants with developmental disabilities.

SPECIFIC AIM 1: To assess the effectiveness of the video-feedback intervention to enhance the socio-emotional behavior of infants with developmental disabilities.

EXPERIMENTAL DESIGN AIM 1: The present research project will include two groups (Video-Feedback Group, VFG; Phone-Call Group, PCG) and four phases: T0, baseline assessment; T1, post-intervention assessment ; T2, follow-up#1 (3 months after the intervention); T3, follow-up#2 (6 months after the intervention). All infants and their mothers will be enrolled at three Child Neuropsychiatric Units in Lombardia Region (OU1, Scientific Institute IRCCS E. Medea; OU2, Fondazione Istituto Neurologico Casimiro Mondino, Pavia, Italy; OU3, Università degli Studi, Brescia, Italy). At each phase, mother-infant interactions will be videotaped during SFP. The VFG dyads will participate to a 6-session videofeedback intervention The aim of the video-feedback intervention is to support maternal sensitivity to the infants' behaviors focusing on different aspects of mother-infant interactions. PCG mothers will be contacted by telephone weekly for 6 weeks, and will be asked for information on their infants' development. No advice about sensitive parenting will be given to the control PCG mothers during these conversations. In each of the three Units, the intervention will be conducted by psychologists/developmental neuropsychiatrists trained on the video-feedback intervention. Infant behavior regulation will be observationally assessed at each of the four phases of the research project.

SPECIFIC AIM 2: To examine the effects of the intervention on maternal responsiveness.

EXPERIMENTAL DESIGN AIM 2: Paralleling infants' behavioral assessment, maternal responsiveness will be assessed at each project phase by means of video-tapes. Additionally, maternal reports of emotional and affective states, including depressive and anxious symptoms and stress perception in taking care of the infant, will be obtained and controlled for. The rate of change over the phases of the project in maternal self-reported emotional states, feelings of attachment and coded sensitivity will concur in defining the efficacy of the intervention in the VFG subjects against the PCG counterparts.

SPECIFIC AIM 3: To investigate the immediate and follow-up pre/post intervention variations in the neuroendocrine functioning (i.e., salivary cortisol and oxytocin) and in the DNA methylation of specific genes associated with infants' behavioral regulation such as: NR3C1, BDNF, SLC6A4, OXTR.

EXPERIMENTAL DESIGN AIM 3: Salivary samples will be collected from the infant at each phase before and after the SFP interaction. For what pertains neuroendocrine markers (i.e., salivary cortisol and oxytocin) saliva will be collected from the infants (and mothers) using an oral cotton swab and it will be collected in eppendorf, centrifuged and conserved according to kit producer guidelines. Samples will be obtained before (1 sample) and after (3 samples: +10, +20, and +30 minutes) the SFP procedure. Due to circadian rhythm of the neuroendocrine systems, all the interactions will occur in the morning, between 9.00 and 12.00 AM. For what pertains the epigenetic profiling, saliva will be collected once per phase. DNA methylation will be assessed at the different CpG sites within the promoter regions of specific target genes (NR3C1, SLC6A4, BDNF, OXTR) previously associated with infants' behavioral development. The rate of change in neuroendocrine concentrations of cortisol and oxytocin as well as the alterations in global and site-specific DNA methylation of the selected genes will be used as independent biomarkers of the effects of the video-feedback intervention.

SIGNIFICANCE AND INNOVATION: First, the study has the potential to bring new evidence in the clinical practices promoting an early intervention for mothers of infants with developmental disabilities. Second, the multi-center nature of this clinical trial will provide a common early intervention program in the Italian context, with potential indirect implication for healthcare costs optimization. Indeed, it has been shown that interventions starting earlier in childhood may be more effective and efficient than those provided in a later period of life. Consistently, the project will be conducted during the first year of life of infants with the potential to permanently alter infants' development trajectories and to yield a significant economic return for the healthcare system. Finally, examining the epigenetic variations related to early parenting intervention the project introduces an innovative approach to early intervention research for families of infants with developmental disabilities.

ELIGIBILITY:
ELIGIBILITY CRITERIA FOR INFANTS

Inclusion Criteria:

* Infants with equivalent age range 3-to-18-months
* Mild to moderate psychomotor delay

Exclusion Criteria:

* Presence of severe sensorial (auditory, visual) deficits
* Genetic syndrome with known functional implications for the epigenetic regulation of target genes

ELIGIBILITY CRITERIA FOR MOTHERS

Inclusion Criteria:

* Mastery of Italian language
* Age > 18 years
* Living with the father of the infant

Exclusion Criteria:

* Documented mental disorder
* Documented disability

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Change in maternal sensitivity | Through study completion: at intervention start (Baseline, T0), 2 months after intervention start (post-intervention, T1), 3 months after intervention end (follow-up, T2), and 6 months after intervention end (follow-up, T3)
  Coded micro-analitically from videotapes of mother-infant interactions.
Change in infant behavioral regulation | Through study completion: at intervention start (Baseline, T0), 2 months after intervention start (post-intervention, T1), 3 months after intervention end (follow-up, T2), and 6 months after intervention end (follow-up, T3)
  Coded micro-analitically from videotapes of mother-infant interactions.

SECONDARY OUTCOMES:
Change in hormones salivary concentrations | Through study completion: at intervention start (Baseline, T0), 2 months after intervention start (post-intervention, T1), 3 months after intervention end (follow-up, T2), and 6 months after intervention end (follow-up, T3)
  Salivary cortisol and oxytocin obtained from infants by trained collaborators.
Change in DNA methylation status | Through study completion: at intervention start (Baseline, T0), 2 months after intervention start (post-intervention, T1), 3 months after intervention end (follow-up, T2), and 6 months after intervention end (follow-up, T3)
  The methylation status of target genes (e.g., NR3C1, SLC6A4, BDNF, OXTR) will be assessed from salivary samples obtained from infants.

OTHER OUTCOMES:
Feasibility and acceptability | Through study completion, 2 months after intervention start (post-intervention, T1)
  Mothers included in the two arms will rate feasibility and acceptability of the respective intervention received.

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Montirosso, PsyD, Principal Investigator — IRCCS E. Medea
Locations (3):
- Italy (3):
  - IRCCS E. Medea, Bosisio Parini, Lecco
  - Università degli Studi di Brescia, Brescia
  - Fondazione Istituto Neurologico Casimiro Mondino, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montirosso R, Rosa E, Giorda R, Fazzi E, Orcesi S, Cavallini A, Provenzi L; Early Intervention Study Group. Early Parenting Intervention - Biobehavioral Outcomes in infants with Neurodevelopmental Disabilities (EPI-BOND): study protocol for an Italian multicentre randomised controlled trial. BMJ Open. 2020 Jul 21;10(7):e035249. doi: 10.1136/bmjopen-2019-035249. PMID 32699128